CLINICAL TRIAL: NCT01545258
Title: Exercise and Changes in Pain Sensitivity in Patients With Knee Osteoarthritis
Brief Title: Exercise and Pain Sensitivity in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Frederiksberg University Hospital (Other)
Responsible Party: Principal Investigator, Marius Henriksen, Senior researcher, Frederiksberg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: PI101.03
Record Dates: First submitted 2012-03-01; First posted 2012-03-06 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-12

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Exercise (Experimental): Exercise training supervised by trained physiotherapists lasting 60 minutes performed 3 times/week.
  Interventions: Other: Exercise
- Control (No Intervention)

INTERVENTIONS:
Other: Exercise — Physiotherapy supervised exercise training. 60 minutes 3 times per week
  Other Names: Exercise training
  Arms: Exercise

SUMMARY:
A commonly administered conservative non-pharmacological treatment for OA is exercise, with beneficial effects in terms of reduced pain and disability.

While the link between exercise and reduced disability is mediated by e.g. increased muscle strength and endurance, the analgesic mechanisms related to exercise are unexplored. knee OA patients have both peripheral and central sensitization of pain mechanisms resulting in hyperalgesia. Thus, targeted pain treatment in these patients may focus on both peripheral and central mechanisms but it unknown if exercise affects either of these mechanisms.

It is hypothesized that in knee OA patients exercise reduces the pain sensitivity

ELIGIBILITY:
Inclusion Criteria:

* Age above 40 years
* Clinical diagnosis of tibiofemoral osteoarthritis
* Radiographic verification of diagnosis (Kellgren&Lawrence 2 or 3)
* Ability to participate in examinations
* Ability to participate in exercise sessions
* 20≤ Body Mass Index (BMI) ≤35 kg/m2
* Ability to comply with rules about concomitant medication and therapy
* Speak, read and write Danish

Exclusion Criteria:

* Participation in exercise training for the knee osteoarthritis within 3 months of enrollment
* Counterindications for exercise
* Pregnant or breastfeeding
* Current or previous autoimmune disease
* History of surgical joint replacement in the lower limbs
* Planned surgery
* Current or previous diagnosis or signs of cardiovascular disease
* Neurological disorders
* Alcohol or drug abuse
* Diabetes
* Psychiatric disorders
* Regional pain syndromes
* Regional pain caused by lumbar or cervical nerve root compression
* Counterindications to MR scan
* Counterindications to MR contrast

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mechanical pain sensitivity | Baseline and at 12 weeks
  Pain thresholds and temporal summation of pain

SECONDARY OUTCOMES:
Change from baseline in proinflammatory cytokines and biomarkers of cartilage breakdown in blood and urine | Baseline and at 12 weeks
Change from baseline in patient reported pain and function | Baseline and at 12 weeks
  KOOS questionnaire
Change from baseline in functional pain test | Baseline and at 12 weeks
  Pain is assessed during continuous tradmill walking at self-selected pace for 20 minutes.
Change from baseline in imaged based quantification of inflammation in the knee | Baseline and at 12 weeks
  Contrast enhanced MRI imaging used to quantify inflammation (DYNAMICA software)

CONTACTS AND LOCATIONS:
Overall Officials: Marius Henriksen, PhD, Principal Investigator — The Parker Institute, Frederiksberg Hospital
Locations (1):
- The Parker Institute, Dept of rheumatology, Frederiksberg hospital, Copenhagen, Denmark

REFERENCES:
- [Derived] Bandak E, Boesen M, Bliddal H, Daugaard C, Hangaard S, Bartholdy C, Damm Nybing J, Kubassova O, Henriksen M. The effect of exercise therapy on inflammatory activity assessed by MRI in knee osteoarthritis: Secondary outcomes from a randomized controlled trial. Knee. 2021 Jan;28:256-265. doi: 10.1016/j.knee.2020.12.022. Epub 2021 Jan 13. PMID 33453514
- [Derived] Bandak E, Boesen M, Bliddal H, Riis RGC, Nielsen SM, Klokker L, Bartholdy C, Nybing JD, Henriksen M. Exercise-induced pain changes associate with changes in muscle perfusion in knee osteoarthritis: exploratory outcome analyses of a randomised controlled trial. BMC Musculoskelet Disord. 2019 Oct 27;20(1):491. doi: 10.1186/s12891-019-2858-8. PMID 31656173
- [Derived] Henriksen M, Klokker L, Bartholdy C, Schjoedt-Jorgensen T, Bandak E, Bliddal H. No effects of functional exercise therapy on walking biomechanics in patients with knee osteoarthritis: exploratory outcome analyses from a randomised trial. BMJ Open Sport Exerc Med. 2017 Mar 27;2(1):e000230. doi: 10.1136/bmjsem-2017-000230. eCollection 2016. PMID 28879038
- [Derived] Bartholdy C, Klokker L, Bandak E, Bliddal H, Henriksen M. A Standardized "Rescue" Exercise Program for Symptomatic Flare-up of Knee Osteoarthritis: Description and Safety Considerations. J Orthop Sports Phys Ther. 2016 Nov;46(11):942-946. doi: 10.2519/jospt.2016.6908. Epub 2016 Sep 28. PMID 27681448
- [Derived] Henriksen M, Klokker L, Graven-Nielsen T, Bartholdy C, Schjodt Jorgensen T, Bandak E, Danneskiold-Samsoe B, Christensen R, Bliddal H. Association of exercise therapy and reduction of pain sensitivity in patients with knee osteoarthritis: a randomized controlled trial. Arthritis Care Res (Hoboken). 2014 Dec;66(12):1836-43. doi: 10.1002/acr.22375. PMID 24905427
- See also: Related Info — http://www.parkerinst.dk